CLINICAL TRIAL: NCT03409315
Title: Prospective Evaluation of impRoving Fluoroquinolone Exposure Using Centralized Tdm in TB Patients
Brief Title: Feasibility of Centralized Therapeutic Drug Monitoring of Fluoroquinolones in Multi-Drug Resistant Tuberculosis Patients
Acronym: PERFECT
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: University Medical Center Groningen (Other)
Responsible Party: Principal Investigator, Jan-Willem C Alffenaar, PhD, PharmD, University Medical Center Groningen
Other Study IDs: CTDM/FQ1
Record Dates: First submitted 2018-01-17; First posted 2018-01-24 (Actual); Last update posted 2019-10-10 (Actual); Status verified 2019-10

CONDITIONS: Tuberculosis, Multidrug-Resistant
Keywords: Centralized Therapeutic Drug Monitoring; Fluoroquinolones
MeSH Terms: conditions — Tuberculosis, Multidrug-Resistant

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (4):
- Moxifloxacin, prospective: Prospective included patients (n=60) receiving centralized therapeutic drug monitoring of moxifloxacin.
  Interventions: Procedure: Centralized Therapeutic Drug Monitoring
- Levofloxacin, prospective: Prospective included patients (n=60) receiving centralized therapeutic drug monitoring of levofloxacin
  Interventions: Procedure: Centralized Therapeutic Drug Monitoring
- Moxifloxacin, historical controls: Historical controls (n=120) matched to prospective patients, did not receive centralized therapeutic drug monitoring of moxifloxacin.
- Levofloxacin, historical controls: Historical controls (n=120) matched to prospective patients, did not receive centralized therapeutic drug monitoring of levofloxacin.

INTERVENTIONS:
Procedure: Centralized Therapeutic Drug Monitoring — Plasma samples will be drawn at peripheral centres en shipped to a central laboratory for analysis. Results and dosing advice will be returned by email to local physician.
  Groups: Levofloxacin, prospective; Moxifloxacin, prospective

SUMMARY:
Observational, multi-centre, prospective study to investigate the feasibility of centralized TDM of moxifloxacin and levofloxacin in MDR-TB patients by determining turn-around time between sampling and receiving dosing advice.

In addition, the effect of TDM will be evaluated by comparing treatment results of prospective patients receiving TDM with historical controls without TDM.

ELIGIBILITY:
Inclusion Criteria:

* Pulmonary MDR-TB
* Sputum smear and sputum culture positive at baseline
* Oral administration of either moxifloxacin or levofloxacin
* Written informed consent (for use of the medical data)

Exclusion Criteria:

* Pregnancy or breast feeding

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Sputum smear and culture positive MDR-TB patients treated with either moxifloxacin or levofloxacin in multiple clinical centres worldwide.
Sampling Method: Probability Sample
Enrollment: 360 (Estimated)
Dates: Start 2018-02-10 (Actual); Primary Completion 2020-11 (Estimated); Study Completion 2020-12 (Estimated)

PRIMARY OUTCOMES:
Feasibility of centralized TDM | 1 week
  Turn-around time between plasma sampling and receiving dosing advice

SECONDARY OUTCOMES:
Impact of centralized TDM | 2 months
  Comparison of % patients with converted sputum smear and culture between prospective patients with TDM and matched historical controls without TDM (1:2)

CONTACTS AND LOCATIONS:
Overall Officials: Jan-WIllem Alffenaar, PhD, Principal Investigator — University Medical Center Groningen
Locations (13):
- The Prince Charles and Caboolture Hospitals, Brisbane, Australia
- Republican Scientific and Practical Centre of Pulmonology and Tuberculosis, Minsk, Belarus
- Hélio Fraga Reference Center, Rio de Janeiro, Brazil
- Athens Chest Hospital "Sotiria", Athens, Greece
- Alma Mater Studiorum University of Bologna, Bologna, Italy
- Reuh Tldc, Upeslejas, Latvia
- Instituto Nacional de Enfermedades Respiratorias, Mexico City, Mexico
- University Medical Center Groningen Beatrixoord, Haren, Netherlands
- Vila Nova Gaia/Espinho Medical School, Vila Nova de Gaia, Portugal
- University of Cape Town, Lung Insitute, Cape Town, South Africa
- Karolinska University Hospital, Stockholm, Sweden
- Kibong'oto Infectious Diseases Hospital, Sanya Juu, Tanzania
- Royal London Hospital, London, United Kingdom

REFERENCES:
- [Derived] van den Elsen SH, Sturkenboom MG, Akkerman O, Barkane L, Bruchfeld J, Eather G, Heysell SK, Hurevich H, Kuksa L, Kunst H, Kuhlin J, Manika K, Moschos C, Mpagama SG, Munoz Torrico M, Skrahina A, Sotgiu G, Tadolini M, Tiberi S, Volpato F, van der Werf TS, Wilson MR, Zuniga J, Touw DJ, Migliori GB, Alffenaar JW. Prospective evaluation of improving fluoroquinolone exposure using centralised therapeutic drug monitoring (TDM) in patients with tuberculosis (PERFECT): a study protocol of a prospective multicentre cohort study. BMJ Open. 2020 Jun 16;10(6):e035350. doi: 10.1136/bmjopen-2019-035350. PMID 32554740